CLINICAL TRIAL: NCT03003468
Title: A Phase Ib/II Study of Anti-PD-1 Antibody Pembrolizumab and Imprime PGG for Patients With Metastatic Non-small Cell Lung Cancer After Progression on First-Line Therapy: Big Ten Cancer Research Consortium BTCRC-LUN15-017
Brief Title: Pembrolizumab + Imprime PGG for Metastatic Non-small Cell Lung Cancer After Progression on First-Line Therapy: Big Ten Cancer Research Consortium BTCRC-LUN15-017
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lawrence Feldman, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); HiberCell, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Feldman, MD, M.D., Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-LUN15-017
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Anti-PD-1; Pembrolizumab; Imprime PGG; MK-3475
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A - Phase Ib (Experimental): Dose Escalation Cohort Cohort 1 will consist of 3-6 patients who will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 2mg/kg on Day 1,8, and 15 of cycles 1-4, and on Day 1 of cycles 5-16. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
  Experimental: Arm A - Phase II Investigational Treatment The maximum safe dose of Imprime PGG in combination with pembrolizumab (as determined in the phase Ib cohort) will be given on Day 1,8, and 15 for cycles 1-4, and on Day 1 of cycles 5-16.
  Cohort 2 will consist of 3-6 patients who will receive pembrolizumab 200mg IV on Day 1 and Imprime PGG at 4mg/kg on Day 1,8, and 15 for Cycles 1-4 and on Day 1 only for Cycles 5-16. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
  Interventions: Drug: Imprime PGG; Drug: MK-3475

INTERVENTIONS:
Drug: Imprime PGG — Arm A: Phase Ib Cohort 1: 2mg/kg IV; Arm A: Phase Ib Cohort 2: 4mg/kg IV
Drug: MK-3475 — 200mg IV
  Other Names: pembrolizumab; Keytruda
Drug: Imprime PGG — Arm B: Phase II treatment: administered at the maximum safe dose of 2mg or 4 mg as established in the Phase Ib cohort study.

SUMMARY:
This is an open label, multi-institutional, single arm study with a dose escalation phase Ib cohort, followed by a phase II cohort of pembrolizumab and Imprime PGG. No randomization or blinding is involved.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

The phase Ib dose escalation will evaluate the combination of pembrolizumab and Imprime PGG for subjects with metastatic non-small cell lung cancer (NSCLC) after progression on first-line platinum-based chemotherapy. The phase II trial will test whether addition of Imprime PGG to pembrolizumab will increase median progression-free survival (PFS) in second line therapy setting in NSCLC.

PHASE Ib DOSE ESCALATION INVESTIGATIONAL TREATMENT:

Cohort 1 will consist of 3-6 patients who will receive

* Imprime PGG 2 mg/kg IV on Days 1, 8, 15 for Cycles 1-4
* Imprime PGG 2 mb/kg IV on Day 1 for Cycles 5-16
* Pembrolizumab 200 mg IV on Day 1 (cycle = 21 days)

Cohort 2 will consist of 3-6 patients who will receive

* Imprime PGG 4 mg/kg IV on Days 1, 8, 15 for Cycles 1-4
* Imprime PGG 2 mb/kg IV on Day 1 for Cycles 5-16
* Pembrolizumab 200 mg IV on Day 1 (cycle = 21 days)

If none of the 3 subjects experience a dose limiting toxicity (DLT) during the first cycle of therapy, an additional three subjects will be enrolled at dose level 2. If all subjects in dose level 2 complete the first cycle of therapy without DLT, 3 more subjects will be enrolled into dose level 2 to ensure only 0-1 of 6 subjects have a DLT. There will be no further escalation beyond dose level 2.

PHASE II INVESTIGATIONAL TREATMENT:

Pembrolizumab will be given on Day 1 of each 21 day cycle after Imprime PGG, and the RP2D dose of Imprime PGG will be given on Days 1, 8 and 15 of each 21 day cycle. Treatment will continue up to 16 cycles, or until disease progression, unacceptable toxicity, subject refusal, or subject death either from progression of disease, the therapy itself, or from other causes.

Life expectancy: of 6 months or greater

The following baseline labs must be completed within 28 days prior to registration for protocol therapy:

Hepatic:

* total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN (except subject with Gilbert's Syndrome, who can have total bilirubin < 3.0 mg/dl)
* aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases

Renal:

* Serum creatinine ≤ 3 mg/dL OR
* if serum creatinine > 3mg/dL, estimated glomerular filtration rate (GFR) ≥ 20 mL/min

Hematopoietic:

* hemoglobin ≥ 9 g/dL, subjects requiring transfusion will not be eligible to start study
* and absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
* and platelet count ≥ 100 × 10^9/L

Coagulation:

* INR < 1.5 × ULN OR
* for subjects receiving anticoagulant, the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for subjects on warfarin should be in the therapeutic range. Low molecular weight heparin (LMWH) is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at time of consent.
* Subjects with histologically or cytologically confirmed non-small cell lung cancer (NCSLC).
* Subjects with stage IV non-small cell lung cancer as defined by American Joint Committee on Cancer (AJCC).
* Phase Ib: Subjects who progressed after first-line platinum-based chemotherapy and who are candidates for second-line therapy.
* Phase II: Subjects who have progressed on first-line systemic therapy (either platinum-based chemotherapy with or without immune checkpoint inhibitor or immune checkpoint inhibitor as first line therapy) who are candidates for second-line systemic therapy. Patients with early stage cancer will also be eligible if progression occurs:

  * within 6 months of adjuvant chemotherapy after curative resection
  * within 6 months of adjuvant chemotherapy after curative resection while on adjuvant immunotherapy, currently only available as part of a clinical trial
  * within 6 months of curative surgery if chemotherapy is given in the neoadjuvant setting
  * within 6 months of completion of chemoradiation (or 6 months from completion of consolidation chemotherapy if administered after concurrent chemoradiation)
  * within 6 months of completion of chemoradiation or consolidation chemotherapy (if administered) while on consolidation immunotherapy, a setting for which durvalumab is FDA approved.
* Phase II: Subjects with an EGFR or ALK mutation who are no longer candidates for TKI therapy and have progressed on standard systemic therapy (either platinum-based chemotherapy with or without immune checkpoint inhibitor or immune checkpoint inhibitor as first line therapy).
* Phase II only: Measurable disease according to RECIST v1.1 (Section 8) obtained by imaging within 28 days prior to study registration. Phase Ib: subjects may enroll with or without measurable disease.
* Phase II only: Subjects must have presence of peripheral blood levels of IgG anti-β-glucan antibody (ABA) of ≥ 20 μg/mL as determined by an ELISA test within 90 days prior to study registration.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 within 28 days prior to study registration.
* Life expectancy of 6 months or greater as determined by the treating physician.
* Adequate hepatic function within 28 days prior to study registration defined as meeting all of the following criteria:

  * total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN (except subject with Gilbert's Syndrome, who can have total bilirubin < 3.0 mg/dl)
  * aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
  * alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* Adequate renal function within 28 days prior to study registration defined by either of the following criteria:

  * Serum creatinine ≤ 3 mg/dL
  * if serum creatinine > 3mg/dL, estimated glomerular filtration rate (GFR) ≥ 20 mL/min
* Adequate hematologic function within 28 days prior to study registration defined as meeting all of the following criteria:

  * hemoglobin ≥ 9 g/dL; subjects requiring transfusion will be eligible to start study
  * and absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * and platelet count ≥ 100 × 109/L
* Adequate coagulation functioning within 28 days prior to study registration defined by either of the following criteria:

  * INR < 1.5 × ULN
  * for subjects receiving anticoagulant, the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for subjects on warfarin should be in the therapeutic range. Low molecular weight heparin (LMWH) is allowed.
* Provided written informed consent and HIPAA authorization for release of personal health information, approved by an Institutional Review Board (IRB). NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Women of childbearing potential (WOCP) must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required within 72 hours of study registration. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required.
* Women of childbearing potential (WOCP) must be willing to use two effective methods of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence for the course of the study until 120 days after the last dose of study drug. NOTE: Women are considered to be of childbearing potential unless they are postmenopausal (≥45 years of age and has not had menses for greater than 12 consecutive months), surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or not heterosexually active for the duration of the study and at least 120 days after the last dose of study drug.
* Men who are not surgically sterile (vasectomy) must agree to use an acceptable method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms from the first dose of study drug through at least 120 days after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.
* Willingness and ability to comply with scheduled visits (including geographical distance), treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Surgery within 4 weeks prior to study registration except for minor procedures. NOTE: Hepatic biliary stent placement, PleurX catheter, port replacement, ureteral stent or other minor surgeries are allowed. NOTE: Subject must have adequately recovered from the toxicity and/or complications of major surgery prior to study registration, as determined by the treating physician.
* Patients with known untreated or active central nervous system (CNS) metastases. Subjects suspected to have brain mets should undergo brain MRI (or CT head if MRI is not feasible) to exclude brain metastases. Patients with treated brain metastases will be eligible as long as their symptoms are improving or achieved new baseline and not requiring steroids for at least 2 weeks. Patients with leptomeningeal disease will be excluded regardless of clinical stability.
* Previously received a solid organ transplant or allogeneic progenitor/stem cell transplant.
* Received a live vaccine within 30 days prior to the first dose of trial treatment. Examples of live vaccines include, but are not limited to: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not allowed.
* History of blood clots, pulmonary embolism, or deep vein thrombosis unless on adequate anticoagulant therapy as determined by the treating investigator (subject must be on stable dose for 2 weeks) and all symptoms have resolved.
* Known history of human immunodeficiency virus [(HIV) HIV 1/2 antibodies].
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Current use of immunosuppressive medication at time of study entry. The following are exceptions to this exclusion criterion: intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection); steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). Cases requiring systemic corticosteroids at physiologic doses must be discussed with Big Ten CRC and HiberCell prior to enrollment.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Exceptions include: patients with controlled diabetes type 1, controlled hypo- or hyperthyroidism, resolved childhood asthma/atopy, vitiligo, or psoriasis not requiring immunosuppressive treatment.
* Received prior chemotherapy, an immune checkpoint inhibitor, or radiation therapy within 2 weeks prior to study registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events from previously administered agents. NOTE: Subjects with alopecia, grade ≤ 2 sensory neuropathy or other grade ≤ 2 AEs not constituting a safety risk based on investigator judgement are an exception to this criterion and can still be considered for the study.
* Any clinically significant infection requiring anti-infective treatment. Patients with infection that is adequately treated will be eligible.
* History of interstitial lung disease requiring immunosuppressive/steroids or history of immunotherapy related pneumonitis that has required steroids or immunosuppression in the past.
* Known history of active tuberculosis.
* Any other severe, uncontrolled medical condition, including uncontrolled diabetes mellitus (defined as a Hemoglobin A1C ≥ 9% in subjects with a prior history of diabetes, 28 days prior to study registration) or unstable congestive heart failure (Stage III-IV of the New York Heart Association Functional Classification).
* Previous known allergy or intolerance to pembrolizumab or any of its excipients.
* Previous exposure or known allergy to Imprime PGG or any of its excipients.
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, interfere with protocol compliance, or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for enrollment in this study.
* Presence of any non-healing wound, fracture, or ulcer within 28 days prior to study registration.
* Any mental or medical condition that prevents the subject from giving informed consent or participating in the trial.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, Gleason ≤ grade 7 prostate cancers, low grade papillary urothelial carcinoma or other cancer for which the subject has been disease-free for at least 2 years. And no additional therapy other than hormonal therapy is required for anticipated to be required during the trial period.
* Treatment with any therapeutic investigational agent within 28 days prior to study registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Feldman, M.D., Study Chair — Big Ten Cancer Research Consortium
Locations (5):
- United States (5):
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Penn State Cancer Institute, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furqan M, Malhotra J, Shergill A, Liu L, Mott SL, Pasquinelli MM, Hulbert A, Kennedy K, Feldman L. Phase Ib/II study of imprime PGG and pembrolizumab in patients with previously treated advanced non-small cell lung cancer (NSCLC): BTCRC LUN 15-017. Transl Lung Cancer Res. 2024 Nov 30;13(11):2998-3009. doi: 10.21037/tlcr-24-346. Epub 2024 Nov 19. PMID 39670007
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase Ib: Imprime PGG 2 mg/kg: Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 2mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
- Phase Ib: Imprime PGG 4 mg/kg: Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 4 mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
- Phase II: Imprime PGG 4 mg/kg: Imprime PGG will be dosed at the dose established as the MTD in Phase Ib (4mg/kg) on Day 1, 8, and 15 for Cycles 1-4, and on Day 1 only for Cycles 5-16 of the 21 day cycle. Pembrolizumab will be infused at 200 mg on Day 1 of the 21 day cycle. On day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab infusion.
Period: Overall Study
Arm/Group | Phase Ib: Imprime PGG 2 mg/kg | Phase Ib: Imprime PGG 4 mg/kg | Phase II: Imprime PGG 4 mg/kg
Started | 3 | 6 | 26
Completed | 3 | 6 | 24
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — No measurable lesions | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: Imprime PGG 2 mg/kg | Phase Ib: Imprime PGG 4 mg/kg | Phase II: Imprime PGG 4 mg/kg | Total
Number analyzed (Participants) | 3 | 6 | 24 | 33
Age, Continuous [Median (Full Range); unit: years] | 68 [66 to 69] | 66 [56 to 72] | 65 [53 to 82] | 66 [53 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 9 | 16
  Male | 1 | 1 | 15 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 5 | 23 | 30
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 7
  White | 1 | 4 | 17 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 24 | 33
Smoking Status [Count of Participants; unit: Participants]
  Never | 0 | 2 | 3 | 5
  Current | 1 | 0 | 6 | 7
  Former | 2 | 4 | 15 | 21
ECOG Performance [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours, and 5=Dead
  Participants
    ECOG = 0 | 0 | 0 | 3 | 3
    ECOG = 1 | 3 | 6 | 20 | 29
    ECOG = 2 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Maximum Tolerated Dose
Description: Phase Ib: Maximum tolerated dose (MTD) for subjects receiving Imprime PGG with pembrolizumab without experiencing dose-limiting toxicity(s) (DLT) per Common Terminology Criteria for Adverse Events (CTCAE) v4.
Time Frame: 21 days
Measure: Number; unit: mg
Groups:
- Phase Ib: Phase Ib (Imprime PGG 2 mg/kg) :
  Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 2mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
  Phase Ib (Imprime PGG 4 mg/kg) :
  Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 4 mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
Arm/Group | Phase Ib
Number analyzed (Participants) | 9
mg
  Imprime PGG | 4
  Pembrolizumab | 200

2. Primary Outcome: Progression Free Survival
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. Progression Free Survival (PFS) is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death. Up to a maximum of 32 months.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint progression-free survival was defined as all patients treated at the MTD, which was determined to be Imprime PGG at 4mg/kg in combination with pembrolizumab 200mg.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Imprime PGG 4 mg/kg: Phase Ib (Imprime PGG 4 mg/kg):
  Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 4 mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
  Phase II (Imprime PGG 4 mg/kg):
  Imprime PGG will be dosed at the dose established as the MTD in Phase Ib (4mg/kg) on Day 1, 8, and 15 for Cycles 1-4, and on Day 1 only for Cycles 5-16 of the 21 day cycle. Pembrolizumab will be infused at 200 mg on Day 1 of the 21 day cycle. On day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab infusion.
Arm/Group | Imprime PGG 4 mg/kg
Number analyzed (Participants) | 30
Months | 2.6 [1.4 to 7]

3. Secondary Outcome: Adverse Events (AEs)
Description: Number of participants with treatment related adverse events regardless of dose are reported by CTCAEv4 term and grade.
Time Frame: AEs have been recorded from the time of consent until 30 days after treatment discontinuation of study drugs or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 13 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for Adverse Events was defined as all patients receiving at least one dose of study treatment regardless of the dosage.
Measure: Count of Participants; unit: Participants
Groups:
- Phase Ib - Phase II: Phase Ib (Imprime PGG 2 mg/kg):
  Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 2mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
  Phase Ib (Imprime PGG 4 mg/kg):
  Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 4 mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
  Phase II (Imprime PGG 4 mg/kg):
  Imprime PGG will be dosed at the dose established as the MTD in Phase Ib (4mg/kg) on Day 1, 8, and 15 for Cycles 1-4, and on Day 1 only for Cycles 5-16 of the 21 day cycle. Pembrolizumab will be infused at 200 mg on Day 1 of the 21 day cycle. On day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab infusion.
Arm/Group | Phase Ib - Phase II
Number analyzed (Participants) | 33
Participants
  Infusion related reaction | 13
  Fatigue / Malaise | 10
  Arthralgia / Myalgia | 7
  Nausea / Vomiting | 7
  Pain | 5
  Rash | 4
  Chills | 3
  Diarrhea | 3
  Dyspnea | 3
  Anorexia | 2
  Cough | 2
  Flu like symptoms | 2
  Headache | 2
  Hypo / Hyperthyroidism | 2
  Pruritus | 2
  Allergic / Injection Site Reaction | 1
  Anemia | 1
  Bloating / Dyspepsia / Flatulence | 1
  Blurred vision | 1
  Colitis | 1
  Creatinine increased | 1
  Dizziness | 1
  Dysphagia | 1
  Fever | 1
  Flushing | 1
  Hyperglycemia | 1
  Hypotension | 1
  Movements involuntary | 1
  Pneumonitis | 1
  Sinus tachycardia | 1

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.The CBR is defined as the proportion of subjects with a confirmed complete response, partial response or stable disease based on RECIST v1.1.
Time Frame: Up to maximum of 32 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Clinical Benefit Rate was defined as all patients treated at the MTD, which was determined to be Imprime PGG at 4mg/kg in combination with pembrolizumab 200mg.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imprime PGG 4 mg/kg
Number analyzed (Participants) | 30
Percentage of participants | 47 [23 to 67]

5. Secondary Outcome: Progression Free Survival (PFS) at 6 Months
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
  PFS at 6 months is defined as the percentage of patient who was progression free at 6 months from the initiation of treatment.
Time Frame: 6 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Progression Free Survival at 6 months was defined as all patients treated at the MTD, which was determined to be Imprime PGG at 4mg/kg in combination with pembrolizumab 200mg.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imprime PGG 4 mg/kg
Number analyzed (Participants) | 30
Percentage of participants | 37 [20 to 55]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: Time of treatment start until death or date of last contact, up to a maximum of 52 months.
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Overall Survival was defined as all patients treated at the MTD, which was determined to be Imprime PGG at 4mg/kg in combination with pembrolizumab 200mg.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imprime PGG 4 mg/kg
Number analyzed (Participants) | 30
Months | 11.1 [7.8 to 18]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 52 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 13 months.
Groups:
- Imprime PGG 2 mg/kg: Phase Ib (Imprime PGG 2 mg/kg):
  Participants will receive pembrolizumab 200mg IV on Day 1 of each 21 day cycle. Imprime PGG will be administered at 2mg/kg on Day 1,8, and 15. On Day 1 of each cycle, the Imprime PGG intravenous infusion is given first followed 15-30 minutes later by the pembrolizumab.
Arm/Group | Imprime PGG 2 mg/kg | Imprime PGG 4 mg/kg
All-Cause Mortality (participants affected / at risk) | 3/3 | 21/30
Serious Adverse Events (participants affected / at risk) | 1/3 | 9/30
Other Adverse Events (participants affected / at risk) | 3/3 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imprime PGG 2 mg/kg (N=3) | Imprime PGG 4 mg/kg (N=30)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
COLITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (2)
INFUSION RELATED REACTION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (2)
NAUSEA (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 2 (3)
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
SEPSIS (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imprime PGG 2 mg/kg (N=3) | Imprime PGG 4 mg/kg (N=30)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 7 (7)
ALLERGIC RHINITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 1 (1)
ANOREXIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 7 (8)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 7 (7)
CHEST WALL PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0)
CHRONIC KIDNEY DISEASE (RENAL AND URINARY DISORDERS) | 1 (1) | 0 (0)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 2 (2) | 5 (5)
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 6 (7)
DEPRESSION (PSYCHIATRIC DISORDERS) | 1 (1) | 2 (2)
DIZZINESS (NERVOUS SYSTEM DISORDERS) | 1 (1) | 4 (4)
DYSPEPSIA (GASTROINTESTINAL DISORDERS) | 1 (1) | 2 (2)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (2) | 5 (11)
EDEMA LIMBS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 3 (3)
ESOPHAGEAL INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 0 (0)
EYE DISORDERS - OTHER, SPECIFY (EYE DISORDERS) | 1 (1) | 0 (0)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 12 (13)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 1 (1) | 1 (1)
GINGIVAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
HEADACHE (NERVOUS SYSTEM DISORDERS) | 2 (4) | 4 (5)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 2 (2)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0)
MYALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 5 (5)
NAUSEA (GASTROINTESTINAL DISORDERS) | 1 (1) | 11 (13)
NEUTROPHIL COUNT DECREASED (INVESTIGATIONS) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 6 (7)
ORAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (5) | 1 (1)
PLATELET COUNT DECREASED (INVESTIGATIONS) | 2 (3) | 0 (0)
PNEUMONITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 1 (1)
PROTEINURIA (RENAL AND URINARY DISORDERS) | 1 (1) | 0 (0)
RECURRENT LARYNGEAL NERVE PALSY (NERVOUS SYSTEM DISORDERS) | 1 (1) | 0 (0)
SINUS PAIN (NERVOUS SYSTEM DISORDERS) | 1 (1) | 0 (0)
SORE THROAT (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 1 (1)
ACUTE KIDNEY INJURY (RENAL AND URINARY DISORDERS) | 0 (0) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (INVESTIGATIONS) | 0 (0) | 1 (1)
ALLERGIC REACTION (IMMUNE SYSTEM DISORDERS) | 0 (0) | 3 (3)
ANEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 (0) | 3 (3)
ANXIETY (PSYCHIATRIC DISORDERS) | 0 (0) | 3 (3)
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 6 (6)
BLOATING (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
BLURRED VISION (EYE DISORDERS) | 0 (0) | 1 (1)
BRONCHOSPASM (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 5 (6)
CONJUNCTIVITIS (EYE DISORDERS) | 0 (0) | 1 (1)
CREATININE INCREASED (INVESTIGATIONS) | 0 (0) | 2 (5)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 0 (0) | 7 (7)
DRY MOUTH (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (1)
DYSPHAGIA (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (EAR AND LABYRINTH DISORDERS) | 0 (0) | 2 (3)
ESOPHAGITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (4)
FLASHING LIGHTS (EYE DISORDERS) | 0 (0) | 1 (2)
FLATULENCE (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (2)
FLU LIKE SYMPTOMS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (2)
FLUSHING (VASCULAR DISORDERS) | 0 (0) | 2 (2)
GAIT DISTURBANCE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
HEARING IMPAIRED (EAR AND LABYRINTH DISORDERS) | 0 (0) | 1 (1)
HEMORRHOIDS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
HOT FLASHES (VASCULAR DISORDERS) | 0 (0) | 1 (1)
HYPERTENSION (VASCULAR DISORDERS) | 0 (0) | 1 (2)
HYPERTHYROIDISM (ENDOCRINE DISORDERS) | 0 (0) | 2 (2)
HYPOMAGNESEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 2 (2)
HYPOTENSION (VASCULAR DISORDERS) | 0 (0) | 1 (1)
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 0 (0) | 2 (2)
INFUSION RELATED REACTION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 11 (21)
INSOMNIA (PSYCHIATRIC DISORDERS) | 0 (0) | 1 (1)
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 3 (3)
LYMPHOCYTE COUNT DECREASED (INVESTIGATIONS) | 0 (0) | 2 (2)
MALAISE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
MOVEMENTS INVOLUNTARY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 1 (1)
NASAL CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (2)
NECK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 2 (2)
OSTEONECROSIS OF JAW (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 1 (1)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (2)
PAIN OF SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (2)
PARESTHESIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PELVIC PAIN (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 2 (3)
PERIPHERAL MOTOR NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
POSTNASAL DRIP (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
PRESYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 2 (2)
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 4 (4)
RASH ACNEIFORM (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 4 (5)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 3 (3)
SINUS TACHYCARDIA (CARDIAC DISORDERS) | 0 (0) | 3 (3)
SINUSITIS (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 3 (3)
SOMNOLENCE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
SYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 0 (0) | 1 (1)
TREMOR (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
TUMOR PAIN (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 2 (3)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 2 (2)
URTICARIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 3 (4)
VAGINAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
VOICE ALTERATION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 2 (2)
VOMITING (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (3)
WEIGHT GAIN (INVESTIGATIONS) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT03003468/Prot_SAP_000.pdf